CLINICAL TRIAL: NCT01647230
Title: Observational Study of Cerebral Oxygenation and Spinal Anaesthesia in Elderly Patients With Hip Fracture
Brief Title: Cerebral Oxygenation and Spinal Anaesthesia in Elderly Patients With Hip Fracture
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital de Sabadell (Other)
Responsible Party: Principal Investigator, Diana L Fernandez Galinski, PhD, Hospital de Sabadell
Other Study IDs: 2011612CSPT
Record Dates: First submitted 2012-07-19; First posted 2012-07-23 (Estimated); Last update posted 2012-07-25 (Estimated); Status verified 2012-07

CONDITIONS: Femoral Fracture; Blood Pressure; Cognitive Impairment
Keywords: Anaesthesia, spinal; Cerebral oximetry; Blood pressure; Heart rate; Cognitive Symptom
MeSH Terms: conditions — Femoral Fractures; Cognitive Dysfunction; Neurobehavioral Manifestations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The aim of this study is to observe how the hemodynamic changes induced by spinal blockade affect cerebral oxygenation. Elderly patients are very frail. Hypotension is very frequent during spinal anaesthesia. Bradycardia is other side effect of regional anaesthesia affecting cardiac output and cerebral blood flow. These complications of spinal anaesthesia could decline cognitive function. In this way a non invasive monitoring technique as cerebral oximetry is useful for the safety of anesthetic procedure.

DETAILED DESCRIPTION:
Patients aged 70 years old with hip fracture presenting for surgical repair under intrathecal anaesthesia performed with bupivacaine or L bupivacaine (dose 7 - 9 mg). Preoperative haemoglobin and drugs consumption are registered. All patients receive supplemental oxygen during surgery. Cerebral oximetry, blood pressure, heart rate and oxygen arterial saturation are measured. Level and duration of sensory and motor block are registered. The study observes if there is any correlation between cerebral oximetry and these hemodynamic parameters.

The investigators also observe if there is any correlation between cerebral oximetry and cognitive function evaluated pre and postoperatively by SPMSQ test.

Postoperative SPMSQ test will be performed on the 5th postoperative day and the complications registered.Patients will be followed for the duration of acute hospital stay.

ELIGIBILITY:
Inclusion criteria:

* Patients aged >70 years old with hip fracture.
* No contraindication for spinal anaesthesia.

Exclusion Criteria:

* Allergic reaction to local anesthetics.
* Severe aortic stenosis.
* Local infection.
* SPMSQ test >7 errors.
* Patient refusal

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients aged > 70 years old with hip fracture undergoing surgery under spinal anaesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2012-02; Study Completion 2013-02 (Estimated)

PRIMARY OUTCOMES:
Cerebral Oximetry | Initial, 3 times after spinal block and every 10 minutes during surgery
  Changes in cerebral oxymetry measured initially (basal), 10, 20 and 30 minutes after spinal block. During surgery oximetry is measured evey 10 minutes to obtain the mean of all the values.
Mean Arterial Pressure (MAP) | Initial, 3 times after spinal block and every 10 minutes during surgery
  Changes in MAP measured initially (basal), 10, 20 and 30 minutes after spinal block. During surgery oximetry is measured every 10 minutes to obtain the mean of all the values
Heart Rate (HR) | Initial, 3 times after spinal block and every 10 minutes during surgery
  Changes in HR (basal), 10, 20 and 30 minutes after spinal block. During surgery oximetry is measured every 10 minutes to obtain the mean of all the values.
Oxygen arterial saturation (OSat) | Initial, 3 times after spinal block and every 10 minutes during surgery
  Changes in OSat measured initially (basal), 10, 20 and 30 minutes after spinal block. During surgery oximetry is measured every 10 minutes to obtain the mean of all the values.

SECONDARY OUTCOMES:
Short Portable Mental Status Questionnaire (SPMSQ) | Once before surgery and at 5th postoperative day
  This test measures cognitive impairment before and after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Diana L Fernández Galinski, PhD, Principal Investigator — Hospital de Sabadell - CSPT
Locations (1):
- Hospital de Sabadell - CSPT, Barcelona, Sabadell, Spain